CLINICAL TRIAL: NCT02195869
Title: A Multicenter Open-Label Phase 1b/2 Study of Ibrutinib in Steroid Dependent or Refractory Chronic Graft Versus Host Disease
Brief Title: Study of the Bruton's Tyrosine Kinase Inhibitor in Subjects With Chronic Graft Versus Host Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-1129-CA
Record Dates: First submitted 2014-07-11; First posted 2014-07-21 (Estimated); Results first posted 2019-07-11 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-06

CONDITIONS: Graft Versus Host Disease
Keywords: PCYC1129; PCYC1129CA; 1129; Ibrutinib; PCI32765; IMBRUVICA; Pharmacyclics; PCYC; GVHD; Steroid dependent; refractory; chronic; graft versus host disease; chronic graft versus host disease; immunology
MeSH Terms: conditions — Graft vs Host Disease; Bronchiolitis Obliterans Syndrome | interventions — ibrutinib

ARMS (4):
- Phase 1b: Dose Level 1 (Experimental): Subjects receive daily dose of 420 mg of Ibrutinib capsules
  Interventions: Drug: Ibrutinib
- Phase 1b: Dose Level 2 (Experimental): Subjects receive daily dose of 280 mg of Ibrutinib capsules
  Interventions: Drug: Ibrutinib
- Phase 1b: Dose Level 3 (Experimental): Subjects receive daily dose of 140 mg of Ibrutinib capsules
  Interventions: Drug: Ibrutinib
- Phase 2 (Experimental): Subjects receive daily dose of recommended phase 2 dose
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Ibrutinib
  Other Names: PCI32765

SUMMARY:
The purpose of this study is to assess the safety and clinical efficacy of ibrutinib in subjects with steroid dependent or refractory Chronic Graft Versus Host Disease.

ELIGIBILITY:
Inclusion Criteria:

* Steroid dependent or refractory classic chronic GVHD disease.
* No more than 3 previous treatments for cGVHD.
* Receiving baseline systemic glucocorticoid therapy (at stable dose) for cGVHD at study entry.
* Men and women ≥18 years old.
* Karnofsky performance status ≥60.

Exclusion Criteria:

* Known or suspected active acute GVHD.
* Current treatment with sirolimus AND either cyclosporine or tacrolimus.
* History of treatment with a tyrosine kinase inhibitor (eg, imatinib), purine analogs or other cancer chemotherapy in the 4 weeks prior to starting study drug.
* Currently active, clinically significant cardiovascular disease.
* Uncontrolled infections not responsive to antibiotics, antiviral medicines, or antifungal medicines or a recent infection requiring systemic treatment that was completed ≤14 days before the first dose of study drug.
* Progressive underlying malignant disease including post-transplant lymphoproliferative disease.
* History of other malignancy (not including the underlying malignancy that was the indication for transplant)
* Concomitant use of warfarin or other Vitamin K antagonists
* Known bleeding disorders or hemophilia.
* History of stroke or intracranial hemorrhage within 6 months prior to enrollment.
* Known history of human immunodeficiency virus (HIV) or active with hepatitis C virus (HCV) or hepatitis B virus (HBV).
* Concurrent use of a strong cytochrome P450(CYP) 3A inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-07-14 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori Styles, MD, Study Director — Pharmacyclics LLC.
Locations (10):
- United States (10):
  - City of Hope Medical Center, Duarte, California
  - University of California, San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - Emory University, Winship Cancer Institute, Atlanta, Georgia
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Vanderbilt University Medical Center, Henry-Joyce Cancer Clinic, Nashville, Tennessee
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

REFERENCES:
- [Derived] Doki N, Toyosaki M, Shiratori S, Osumi T, Okada M, Kawakita T, Sawa M, Ishikawa T, Ueda Y, Yoshinari N, Nakahara S. An Open-Label, Single-Arm, Multicenter Study of Ibrutinib in Japanese Patients With Steroid-dependent/Refractory Chronic Graft-Versus-Host Disease. Transplant Cell Ther. 2021 Oct;27(10):867.e1-867.e9. doi: 10.1016/j.jtct.2021.05.019. Epub 2021 Jun 6. PMID 34102349
- [Derived] Waller EK, Miklos D, Cutler C, Arora M, Jagasia MH, Pusic I, Flowers MED, Logan AC, Nakamura R, Chang S, Clow F, Lal ID, Styles L, Jaglowski S. Ibrutinib for Chronic Graft-versus-Host Disease After Failure of Prior Therapy: 1-Year Update of a Phase 1b/2 Study. Biol Blood Marrow Transplant. 2019 Oct;25(10):2002-2007. doi: 10.1016/j.bbmt.2019.06.023. Epub 2019 Jun 28. PMID 31260802
- [Derived] Miklos D, Cutler CS, Arora M, Waller EK, Jagasia M, Pusic I, Flowers ME, Logan AC, Nakamura R, Blazar BR, Li Y, Chang S, Lal I, Dubovsky J, James DF, Styles L, Jaglowski S. Ibrutinib for chronic graft-versus-host disease after failure of prior therapy. Blood. 2017 Nov 23;130(21):2243-2250. doi: 10.1182/blood-2017-07-793786. Epub 2017 Sep 18. PMID 28924018

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1b/Phase 2: Subjects receive daily dose of 420 mg of Ibrutinib capsules
Period: Overall Study
Arm/Group | Phase 1b/Phase 2
Started | 42 (Phase 1b: 6 patients, 420 mg, no DLT observed. Phase 2: 42 patients, 420 mg)
All-Treated Population | 42
Completed | 0
Not Completed | 42
Not completed — cGVHD Progression | 5
Not completed — Malignancy Progression/relapse | 2
Not completed — Adverse Event | 15
Not completed — Withdrawal by Subject | 7
Not completed — Physician Decision | 4
Not completed — Study Terminated by Sponsor | 7
Not completed — Noncompliance with study drug | 2

BASELINE CHARACTERISTICS:
Population: Baseline analysis population includes all participants that received at least 1 dose of ibrutinib.
Arm/Group | Phase 1b/Phase 2
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.5 (15.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 39
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: To Evaluate the Safety and Tolerability of Ibrutinib in Steroid Dependent/Refractory cGVHD.
Description: Number of participants with dose-limiting toxicities as a measure of safety profile to determine recommended dose of ibrutinib
Time Frame: 28 treatment days after last subject enrolled in Phase 1 dose level(s).
Population: Endpoint only includes Phase 1 data.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1b: Dose Level 1: Subjects receive daily dose of 420 mg of Ibrutinib capsules for dose level 1
- Phase 2: Subjects receive daily dose of 420 mg of Ibrutinib capsules
Arm/Group | Phase 1b: Dose Level 1 | Phase 2
Number analyzed (Participants) | 6 | 0
Participants | 0 |

2. Primary Outcome: Phase 2: Overall Response Rate as the Percentage of Participants With Response
Description: Overall Response Rate is defined as the proportion of subjects who achieved complete response (CR) or partial response (PR). Response criteria are based on NIH cGVHD Response assessment (Pavletic 2006; Measurement of Therapeutic Response, ASBMT Web site).
Time Frame: Analysis was conducted with the data extraction date of 15 Sep 2017, with a median follow-up time of 25.56 months.
Population: Efficacy analyses were performed using the All-treated Population (N = 42)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase1b/Phase 2: Subjects receive daily dose of 420 mg of Ibrutinib capsules
Arm/Group | Phase1b/Phase 2
Number analyzed (Participants) | 42
percentage of participants | 69 [52.9 to 82.4]

3. Secondary Outcome: Sustained Response Rate as the Percentage of Participants With Sustained Response
Description: For subjects who achieved an NIH-defined CR or PR, the proportion of subjects who achieved CR or PR that was sustained for at least 20 weeks (140 days). Intermittent SD was also acceptable.
Time Frame: Analysis was conducted with the data extraction date of 15 Sep 2017, with a median follow-up time of 25.56 months.
Population: Phase 2 subjects include all subjects who participated in phase 1b. Subjects evaluated for sustained response includes participants who had achieved an NIH-defined CR or PR.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase1b/Phase 2
Number analyzed (Participants) | 29
percentage of participants | 69 [49.2 to 84.7]

4. Secondary Outcome: To Evaluate the Clinical Efficacy of Ibrutinib in Steroid Dependent/Refractory cGVHD by Measuring: Duration of Response (DOR)
Description: For subjects who achieved an NIH-defined CR or PR, the interval between the date of initial documentation of a response and the date of first documented evidence of PD, death, or date of censoring if applicable.
Time Frame: Analysis was conducted with the data extraction date of 15 Sep 2017, with a median follow-up time of 25.56 months.
Population: Phase 2 subjects includes all subjects who participated in Phase 1b
Measure: Median (95% Confidence Interval); unit: Median
Arm/Group | Phase1b/Phase 2
Number analyzed (Participants) | 29
Median | NA [NA to NA] — NA means not achieved or not estimable.

5. Secondary Outcome: Corticosteroid Requirement Changes Over Time
Description: Average daily corticosteroid dose assessed each week.
Time Frame: Analysis was conducted with the data extraction date of 15 Sep 2017, with a median follow-up time of 25.56 months.
Population: Phase 2 subjects includes all subjects who participated in Phase 1b.
Measure: Median (Full Range); unit: Daily Dose of Steroid by Weight (mg/kg/d
Arm/Group | Phase 1b/Phase 2
Number analyzed (Participants) | 42
Daily Dose of Steroid by Weight (mg/kg/d
  Week 1 | 0.31 [0.06 to 1.3]
  Week 2 | 0.32 [0.06 to 1.35]
  Week 3 | 0.32 [0.06 to 1.35]
  Week 4: number analyzed (Participants) | 41
  Week 4 | 0.31 [0.06 to 1.35]
  Week 5: number analyzed (Participants) | 41
  Week 5 | 0.31 [0.06 to 1.53]
  Week 6: number analyzed (Participants) | 41
  Week 6 | 0.30 [0.06 to 1.53]
  Week 7: number analyzed (Participants) | 41
  Week 7 | 0.30 [0.06 to 1.53]
  Week 8: number analyzed (Participants) | 39
  Week 8 | 0.30 [0.01 to 1.53]
  Week 9: number analyzed (Participants) | 37
  Week 9 | 0.27 [0.00 to 1.03]
  Week 10: number analyzed (Participants) | 36
  Week 10 | 0.25 [0.00 to 1.54]
  Week 11: number analyzed (Participants) | 33
  Week 11 | 0.25 [0.00 to 2.02]
  Week 12: number analyzed (Participants) | 30
  Week 12 | 0.25 [0.00 to 0.62]
  Week 13: number analyzed (Participants) | 29
  Week 13 | 0.24 [0.00 to 0.62]
  Week 14: number analyzed (Participants) | 28
  Week 14 | 0.23 [0.00 to 0.57]
  Week 15: number analyzed (Participants) | 28
  Week 15 | 0.23 [0.00 to 0.58]
  Week 16: number analyzed (Participants) | 27
  Week 16 | 0.23 [0.00 to 0.48]
  Week 17: number analyzed (Participants) | 26
  Week 17 | 0.21 [0.00 to 0.47]
  Week 18: number analyzed (Participants) | 26
  Week 18 | 0.20 [0.00 to 0.44]
  Week 19: number analyzed (Participants) | 26
  Week 19 | 0.20 [0.00 to 0.44]
  Week 20: number analyzed (Participants) | 26
  Week 20 | 0.21 [0.00 to 0.44]
  Week 21: number analyzed (Participants) | 26
  Week 21 | 0.22 [0.00 to 0.37]
  Week 22: number analyzed (Participants) | 26
  Week 22 | 0.22 [0.00 to 0.37]
  Week 23: number analyzed (Participants) | 26
  Week 23 | 0.22 [0.00 to 0.60]
  Week 24: number analyzed (Participants) | 26
  Week 24 | 0.21 [0.00 to 0.37]
  Week 25: number analyzed (Participants) | 26
  Week 25 | 0.19 [0.00 to 0.38]
  Week 26: number analyzed (Participants) | 23
  Week 26 | 0.18 [0.00 to 0.37]
  Week 27: number analyzed (Participants) | 23
  Week 27 | 0.18 [0.00 to 0.37]
  Week 28: number analyzed (Participants) | 23
  Week 28 | 0.18 [0.00 to 0.37]
  Week 29: number analyzed (Participants) | 23
  Week 29 | 0.16 [0.00 to 0.37]
  Week 30: number analyzed (Participants) | 23
  Week 30 | 0.16 [0.00 to 0.32]
  Week 31: number analyzed (Participants) | 23
  Week 31 | 0.16 [0.00 to 0.29]
  Week 32: number analyzed (Participants) | 22
  Week 32 | 0.18 [0.00 to 0.29]
  Week 33: number analyzed (Participants) | 22
  Week 33 | 0.17 [0.00 to 0.29]
  Week 34: number analyzed (Participants) | 22
  Week 34 | 0.17 [0.00 to 0.29]
  Week 35: number analyzed (Participants) | 21
  Week 35 | 0.18 [0.00 to 0.29]
  Week 36: number analyzed (Participants) | 21
  Week 36 | 0.18 [0.00 to 0.29]
  Week 37: number analyzed (Participants) | 21
  Week 37 | 0.16 [0.00 to 0.29]
  Week 38: number analyzed (Participants) | 21
  Week 38 | 0.15 [0.00 to 0.35]
  Week 39: number analyzed (Participants) | 20
  Week 39 | 0.15 [0.00 to 0.30]
  Week 40: number analyzed (Participants) | 20
  Week 40 | 0.15 [0.00 to 0.30]
  Week 41: number analyzed (Participants) | 20
  Week 41 | 0.15 [0.00 to 0.30]
  Week 42: number analyzed (Participants) | 20
  Week 42 | 0.15 [0.00 to 0.30]
  Week 43: number analyzed (Participants) | 20
  Week 43 | 0.13 [0.00 to 0.30]
  Week 44: number analyzed (Participants) | 20
  Week 44 | 0.13 [0.00 to 0.21]
  Week 45: number analyzed (Participants) | 20
  Week 45 | 0.13 [0.00 to 0.21]
  Week 46: number analyzed (Participants) | 19
  Week 46 | 0.13 [0.00 to 0.60]
  Week 47: number analyzed (Participants) | 19
  Week 47 | 0.13 [0.00 to 0.60]
  Week 48: number analyzed (Participants) | 19
  Week 48 | 0.13 [0.00 to 0.53]
  Week 49: number analyzed (Participants) | 19
  Week 49 | 0.12 [0.00 to 0.46]
  Week 50: number analyzed (Participants) | 19
  Week 50 | 0.10 [0.00 to 0.36]
  Week 51: number analyzed (Participants) | 19
  Week 51 | 0.10 [0.00 to 0.24]
  Week 52: number analyzed (Participants) | 19
  Week 52 | 0.10 [0.00 to 0.24]
  Week 53: number analyzed (Participants) | 19
  Week 53 | 0.10 [0.00 to 0.24]
  Week 54: number analyzed (Participants) | 19
  Week 54 | 0.10 [0.00 to 0.24]
  Week 55: number analyzed (Participants) | 19
  Week 55 | 0.10 [0.00 to 0.24]
  Week 56: number analyzed (Participants) | 19
  Week 56 | 0.10 [0.00 to 0.24]
  Week 57: number analyzed (Participants) | 19
  Week 57 | 0.10 [0.00 to 0.24]
  Week 58: number analyzed (Participants) | 18
  Week 58 | 0.10 [0.00 to 0.21]
  Week 59: number analyzed (Participants) | 18
  Week 59 | 0.10 [0.00 to 0.27]
  Week 60: number analyzed (Participants) | 18
  Week 60 | 0.08 [0.00 to 0.21]
  Week 61: number analyzed (Participants) | 18
  Week 61 | 0.08 [0.00 to 0.21]
  Week 62: number analyzed (Participants) | 16
  Week 62 | 0.08 [0.00 to 0.21]
  Week 63: number analyzed (Participants) | 16
  Week 63 | 0.08 [0.00 to 0.21]
  Week 64: number analyzed (Participants) | 16
  Week 64 | 0.08 [0.00 to 0.21]
  Week 65: number analyzed (Participants) | 16
  Week 65 | 0.08 [0.00 to 0.21]
  Week 66: number analyzed (Participants) | 16
  Week 66 | 0.08 [0.00 to 0.21]
  Week 67: number analyzed (Participants) | 16
  Week 67 | 0.08 [0.00 to 0.21]
  Week 68: number analyzed (Participants) | 16
  Week 68 | 0.08 [0.00 to 0.21]
  Week 69: number analyzed (Participants) | 16
  Week 69 | 0.08 [0.00 to 0.21]
  Week 70: number analyzed (Participants) | 15
  Week 70 | 0.08 [0.00 to 0.21]
  Week 71: number analyzed (Participants) | 15
  Week 71 | 0.07 [0.00 to 0.21]
  Week 72: number analyzed (Participants) | 15
  Week 72 | 0.08 [0.00 to 0.21]
  Week 73: number analyzed (Participants) | 15
  Week 73 | 0.08 [0.00 to 0.21]
  Week 74: number analyzed (Participants) | 14
  Week 74 | 0.07 [0.00 to 0.21]
  Week 75: number analyzed (Participants) | 14
  Week 75 | 0.07 [0.00 to 0.20]
  Week 76: number analyzed (Participants) | 14
  Week 76 | 0.07 [0.00 to 0.20]
  Week 77: number analyzed (Participants) | 14
  Week 77 | 0.07 [0.00 to 0.20]
  Week 78: number analyzed (Participants) | 14
  Week 78 | 0.07 [0.00 to 0.20]
  Week 79: number analyzed (Participants) | 14
  Week 79 | 0.07 [0.00 to 0.20]
  Week 80: number analyzed (Participants) | 14
  Week 80 | 0.07 [0.00 to 0.20]
  Week 81: number analyzed (Participants) | 14
  Week 81 | 0.07 [0.00 to 0.27]
  Week 82: number analyzed (Participants) | 14
  Week 82 | 0.07 [0.00 to 0.31]
  Week 83: number analyzed (Participants) | 14
  Week 83 | 0.07 [0.00 to 0.31]
  Week 84: number analyzed (Participants) | 13
  Week 84 | 0.07 [0.00 to 0.31]
  Week 85: number analyzed (Participants) | 12
  Week 85 | 0.08 [0.00 to 0.31]
  Week 86: number analyzed (Participants) | 12
  Week 86 | 0.08 [0.00 to 0.32]
  Week 87: number analyzed (Participants) | 12
  Week 87 | 0.08 [0.00 to 0.32]
  Week 88: number analyzed (Participants) | 12
  Week 88 | 0.08 [0.00 to 0.32]
  Week 89: number analyzed (Participants) | 12
  Week 89 | 0.08 [0.00 to 0.95]
  Week 90: number analyzed (Participants) | 12
  Week 90 | 0.08 [0.00 to 0.95]
  Week 91: number analyzed (Participants) | 12
  Week 91 | 0.08 [0.00 to 0.95]
  Week 92: number analyzed (Participants) | 12
  Week 92 | 0.08 [0.00 to 0.95]
  Week 93: number analyzed (Participants) | 12
  Week 93 | 0.08 [0.00 to 0.95]
  Week 94: number analyzed (Participants) | 12
  Week 94 | 0.08 [0.00 to 0.95]
  Week 95: number analyzed (Participants) | 11
  Week 95 | 0.08 [0.00 to 0.95]
  Week 96: number analyzed (Participants) | 11
  Week 96 | 0.08 [0.00 to 0.95]
  Week 97: number analyzed (Participants) | 11
  Week 97 | 0.08 [0.00 to 0.95]
  Week 98: number analyzed (Participants) | 11
  Week 98 | 0.08 [0.00 to 0.95]
  Week 99: number analyzed (Participants) | 11
  Week 99 | 0.08 [0.00 to 0.95]
  Week 100: number analyzed (Participants) | 11
  Week 100 | 0.08 [0.00 to 0.95]
  Week 101: number analyzed (Participants) | 11
  Week 101 | 0.09 [0.00 to 0.95]
  Week 102: number analyzed (Participants) | 11
  Week 102 | 0.09 [0.00 to 0.95]
  Week 103: number analyzed (Participants) | 11
  Week 103 | 0.09 [0.00 to 0.95]
  Week 104: number analyzed (Participants) | 11
  Week 104 | 0.09 [0.00 to 0.95]
  Week 105: number analyzed (Participants) | 11
  Week 105 | 0.08 [0.00 to 0.95]
  Week 106: number analyzed (Participants) | 11
  Week 106 | 0.08 [0.00 to 0.95]
  Week 107: number analyzed (Participants) | 11
  Week 107 | 0.08 [0.00 to 0.95]
  Week 108: number analyzed (Participants) | 11
  Week 108 | 0.08 [0.00 to 0.95]
  Week 109: number analyzed (Participants) | 11
  Week 109 | 0.08 [0.00 to 0.95]
  Week 110: number analyzed (Participants) | 11
  Week 110 | 0.08 [0.00 to 0.95]
  Week 111: number analyzed (Participants) | 11
  Week 111 | 0.08 [0.00 to 0.95]
  Week 112: number analyzed (Participants) | 9
  Week 112 | 0.08 [0.00 to 0.95]
  Week 113: number analyzed (Participants) | 8
  Week 113 | 0.08 [0.00 to 0.95]
  Week 114: number analyzed (Participants) | 8
  Week 114 | 0.08 [0.00 to 0.95]
  Week 115: number analyzed (Participants) | 8
  Week 115 | 0.12 [0.00 to 0.95]
  Week 116: number analyzed (Participants) | 8
  Week 116 | 0.12 [0.00 to 0.95]
  Week 117: number analyzed (Participants) | 7
  Week 117 | 0.08 [0.00 to 0.95]
  Week 118: number analyzed (Participants) | 7
  Week 118 | 0.08 [0.00 to 0.95]
  Week 119: number analyzed (Participants) | 7
  Week 119 | 0.08 [0.00 to 0.95]
  Week 120: number analyzed (Participants) | 7
  Week 120 | 0.08 [0.00 to 0.95]
  Week 121: number analyzed (Participants) | 7
  Week 121 | 0.08 [0.00 to 0.95]
  Week 122: number analyzed (Participants) | 6
  Week 122 | 0.12 [0.00 to 0.95]
  Week 123: number analyzed (Participants) | 5
  Week 123 | 0.08 [0.00 to 0.22]
  Week 124: number analyzed (Participants) | 5
  Week 124 | 0.08 [0.00 to 0.22]
  Week 125: number analyzed (Participants) | 5
  Week 125 | 0.08 [0.00 to 0.22]
  Week 126: number analyzed (Participants) | 4
  Week 126 | 0.08 [0.00 to 0.22]
  Week 127: number analyzed (Participants) | 4
  Week 127 | 0.08 [0.00 to 0.22]
  Week 128: number analyzed (Participants) | 3
  Week 128 | 0.00 [0.00 to 0.22]
  Week 129: number analyzed (Participants) | 3
  Week 129 | 0.00 [0.00 to 0.22]
  Week 130: number analyzed (Participants) | 3
  Week 130 | 0.00 [0.00 to 0.22]
  Week 131: number analyzed (Participants) | 3
  Week 131 | 0.00 [0.00 to 0.19]
  Week 132: number analyzed (Participants) | 3
  Week 132 | 0.00 [0.00 to 0.15]
  Week 133: number analyzed (Participants) | 3
  Week 133 | 0.00 [0.00 to 0.15]
  Week 134: number analyzed (Participants) | 3
  Week 134 | 0.00 [0.00 to 0.15]
  Week 135: number analyzed (Participants) | 3
  Week 135 | 0.00 [0.00 to 0.15]
  Week 136: number analyzed (Participants) | 3
  Week 136 | 0.00 [0.00 to 0.15]
  Week 137: number analyzed (Participants) | 3
  Week 137 | 0.00 [0.00 to 0.15]
  Week 138: number analyzed (Participants) | 3
  Week 138 | 0.00 [0.00 to 0.15]
  Week 139: number analyzed (Participants) | 3
  Week 139 | 0.00 [0.00 to 0.15]
  Week 140: number analyzed (Participants) | 3
  Week 140 | 0.00 [0.00 to 0.15]
  Week 141: number analyzed (Participants) | 3
  Week 141 | 0.00 [0.00 to 0.16]
  Week 142: number analyzed (Participants) | 3
  Week 142 | 0.00 [0.00 to 0.17]
  Week 143: number analyzed (Participants) | 3
  Week 143 | 0.00 [0.00 to 0.17]
  Week 144: number analyzed (Participants) | 3
  Week 144 | 0.00 [0.00 to 0.17]
  Week 145: number analyzed (Participants) | 3
  Week 145 | 0.00 [0.00 to 0.17]
  Week 146: number analyzed (Participants) | 3
  Week 146 | 0.00 [0.00 to 0.17]
  Week 147: number analyzed (Participants) | 3
  Week 147 | 0.00 [0.00 to 0.17]
  Week 148: number analyzed (Participants) | 3
  Week 148 | 0.00 [0.00 to 0.17]
  Week 149: number analyzed (Participants) | 3
  Week 149 | 0.00 [0.00 to 0.17]
  Week 150: number analyzed (Participants) | 3
  Week 150 | 0.00 [0.00 to 0.17]
  Week 151: number analyzed (Participants) | 3
  Week 151 | 0.00 [0.00 to 0.17]
  Week 152: number analyzed (Participants) | 3
  Week 152 | 0.00 [0.00 to 0.17]
  Week 153: number analyzed (Participants) | 3
  Week 153 | 0.00 [0.00 to 0.15]
  Week 154: number analyzed (Participants) | 3
  Week 154 | 0.00 [0.00 to 0.14]
  Week 155: number analyzed (Participants) | 3
  Week 155 | 0.00 [0.00 to 0.14]
  Week 156: number analyzed (Participants) | 3
  Week 156 | 0.00 [0.00 to 0.14]
  Week 157: number analyzed (Participants) | 3
  Week 157 | 0.00 [0.00 to 0.13]
  Week 158: number analyzed (Participants) | 2
  Week 158 | 0.06 [0.00 to 0.11]
  Week 159: number analyzed (Participants) | 2
  Week 159 | 0.06 [0.00 to 0.11]
  Week 160: number analyzed (Participants) | 2
  Week 160 | 0.06 [0.00 to 0.11]

6. Secondary Outcome: Percentage of Participants With Overall Improvement in Lee cGVHD Symptom Summary Score
Description: Subject reported improvement in symptom burden. The symptom burden will be measured according to the Lee cGVHD Symptom Scale. A change in >7 points on the Lee cGVHD Symptom Scale will be considered significant and relates to improvement in quality of life.
  A score is calculated for each subscale by taking the mean of all items completed if more than 50% were answered and normalizing to a 0 to 100 scale. A total summary score is calculated as the average of these 7 subscales if at least 4 subscales have valid scores.
  There are 7 subscales (Skin, Energy, Lung, Eye, Nutrition, Mouth and Psychological) with ratings as follow: 0- Not at all, 1- Slightly, 2 Moderately, 3 Quite a bit, 4-Extremely; with a lower values representing a better outcome.
Time Frame: Analysis was conducted with the data extraction date of 15 Sep 2017, with a median follow-up time of 25.56 months.
Population: All subjects who received at least 1 dose of ibrutinib at the recommended Phase 2 dose.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1b/Phase 2
Number analyzed (Participants) | 42
percentage of participants | 42.9 [27.7 to 59]

7. Secondary Outcome: Phase 2b: To Evaluate the Safety and Tolerability of Ibrutinib in Steroid Dependent/Refractory cGVHD
Description: Number of Participants With Adverse Events as a Measure of Safety and Tolerability of Ibrutinib
Time Frame: From first dose with study drug until 30 days after the last dose of study drug, up to 36.7 months
Population: Phase 2 subjects includes all subjects who participated in Phase 1b
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b/Phase 2
Number analyzed (Participants) | 42
Participants | 42

ADVERSE EVENTS:
Time Frame: From first dose of study drug to within 30 days of last dose or starting subsequent therapy for cGVHD, up to 36.7 months
Description: Adverse events were not collected by phase because the phase 1 part of the study confirmed the first dose level (420mg was acceptable for cGVHD subjects and it was used as the recommended Phase 2 dose (RP2D). The Safety Population was the same as the All-treated Population (ie, all subject who received at least 1 dose of ibrutinib at the RP2D)
Arm/Group | Phase1b/Phase 2
All-Cause Mortality (participants affected / at risk) | 7/42
Serious Adverse Events (participants affected / at risk) | 22/42
Other Adverse Events (participants affected / at risk) | 41/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase1b/Phase 2 (N=42)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 6
Cellulitis (Infections and infestations) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Headache (Nervous system disorders) | 2
Septic shock (Infections and infestations) | 2
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Atrial fibrilation (Cardiac disorders) | 1
Bacteraemia (Infections and infestations) | 1
Brain abscess (Infections and infestations) | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 1
Clostridium difficile infection (Infections and infestations) | 1
Compression fracture (Injury, poisoning and procedural complications) | 1
Deep vein thrombosis (Vascular disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Electrocardiogram QT prolonged (Investigations) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Graft versus host disease (Immune system disorders) | 1
Hypertension (Vascular disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Pneumonia viral (Infections and infestations) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Prolymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pyrexia (General disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Rhinovirus infection (Infections and infestations) | 1
Skin mass (Skin and subcutaneous tissue disorders) | 1
Staphylococcal bacteraemia (Infections and infestations) | 1
Syncope (Nervous system disorders) | 1
Urinary tract infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase1b/Phase 2 (N=42)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 17
Increased tendency to bruise (Blood and lymphatic system disorders) | 10
Anaemia (Blood and lymphatic system disorders) | 3
Cardiac Disorders (Cardiac disorders) | 11
Sinus tachycardia (Cardiac disorders) | 4
Tachycardia (Cardiac disorders) | 3
Eye disorders (Eye disorders) | 11
Gastrointestinal disorders (Gastrointestinal disorders) | 38
Diarrhoea (Gastrointestinal disorders) | 17
Nausea (Gastrointestinal disorders) | 12
Constipation (Gastrointestinal disorders) | 5
Mouth Ulceration (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 5
Abdominal Pain (Gastrointestinal disorders) | 4
Dry mouth (Gastrointestinal disorders) | 4
Gastroesophogeal reflux disease (Gastrointestinal disorders) | 4
Dysphagia (Gastrointestinal disorders) | 3
Oral pain (Gastrointestinal disorders) | 3
Stomatitis (Gastrointestinal disorders) | 3
General disorders and administration site conditions (General disorders) | 30
Fatique (General disorders) | 24
Pyrexia (General disorders) | 7
Oedema peripheral (General disorders) | 6
Influenza like illness (General disorders) | 3
Hepatobiliary disorders (Hepatobiliary disorders) | 4
Hepatic function abnormal (Hepatobiliary disorders) | 4
Immune system disorders (Immune system disorders) | 6
Infections and infestations (Infections and infestations) | 25
Upper respiratory tract infection (Infections and infestations) | 8
Cellulitis (Infections and infestations) | 4
Cytomegalovirus infection (Infections and infestations) | 3
Urinary tract infections (Infections and infestations) | 3
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 14
Fall (Injury, poisoning and procedural complications) | 7
Contusion (Injury, poisoning and procedural complications) | 5
Laceration (Injury, poisoning and procedural complications) | 3
Investigations (Investigations) | 10
Weight decreased (Investigations) | 4
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 16
Hyperglycaemia (Metabolism and nutrition disorders) | 5
Hypokalaemia (Metabolism and nutrition disorders) | 5
Hypophosphataemia (Metabolism and nutrition disorders) | 5
Decreased appetite (Metabolism and nutrition disorders) | 4
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 20
Muscle spasms (Musculoskeletal and connective tissue disorders) | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Neoplasms benign, malignant unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Nervous system disorders (Nervous system disorders) | 17
Headache (Nervous system disorders) | 7
Dizziness (Nervous system disorders) | 4
Somnolence (Nervous system disorders) | 3
Psychiatric disorders (Psychiatric disorders) | 12
Anxiety (Psychiatric disorders) | 4
Delerium (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 3
Renal and urinary disorders (Renal and urinary disorders) | 5
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 18
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 19
Night Sweats (Skin and subcutaneous tissue disorders) | 3
Vascular disorders (Vascular disorders) | 9
Hypertension (Vascular disorders) | 3
Hypotension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution/Investigator will not publish without Sponsor prior review and approval.

DOCUMENTS (2):
  • Study Protocol (2015-10-21): https://cdn.clinicaltrials.gov/large-docs/69/NCT02195869/Prot_000.pdf
  • Statistical Analysis Plan (2016-08-31): https://cdn.clinicaltrials.gov/large-docs/69/NCT02195869/SAP_001.pdf